CLINICAL TRIAL: NCT00380679
Title: Offering Influenza and Pneumococcal Vaccine to Patients Being Evaluated in the Emergency Department
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5800
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2006-09-26 (Estimated); Status verified 2006-09

CONDITIONS: High Risk for Serious Influenza; High Risk for Pneumonia
MeSH Terms: interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza vaccination
Biological: Pneumococcal polysaccharide vaccination

SUMMARY:
According to the Advisory Committee on Immunization Practices (ACIP), all people aged 50 years or older and persons aged less than 50 years who have medical conditions that put them at increased risk for serious influenza disease should receive an annual influenza vaccination. However, since the mid-1990s, vaccination rates and racial disparities have mostly remained static, and there has been limited progress towards the Healthy People 2010 objectives for influenza vaccination coverage.

The purpose of this study is to determine what proportion of previously unvaccinated persons in target groups for whom influenza and pneumococcal vaccine are recommended will accept and receive influenza and/or pneumococcal vaccine in an urban emergency department (ED), and to estimate the potential impact of ED vaccination on population-based vaccination coverage. The intervention will utilize a combination of assessment survey, vaccine information and pre-printed vaccine order sheets.

The target population for influenza vaccinations includes all patients aged 18 years and older for whom influenza vaccine is recommended by the ACIP. This includes all persons aged 50 years and older and persons aged 18 to 49 years who are in one of the following groups: 1) health care workers, 2) pregnant women, 3) residents of long-term care facilities, 4) household contacts and out-of-home caregivers of children aged 0 to 23 months, or 5) persons with underlying chronic medical conditions which increase their risk of influenza-related complications. The target population for pneumococcal vaccination includes all patients aged 65 years or older who have not previously been vaccinated against pneumococcus or have not received the vaccine within 5 years (and were less than 65 years at the time of vaccination).

DETAILED DESCRIPTION:
PROTOCOL - Baton Rouge General Medical Center

Background

According to the Institute of Medicine, non-institutionalized high-risk adults may present the greatest challenge to adult immunizations. There are a number of barriers to implementation of comprehensive strategies for vaccinating adults:

* Routine preventive health visits are infrequent and transient
* Individuals lack knowledge of the vaccines required during adulthood
* Primary care providers may lack time, knowledge, or ability to perform a vaccination assessment, or it may not be part of their standard practice pattern
* Primary care providers lack the infrastructure (especially time and personnel) to assist with adequately assessing and documenting immunization status

Emergency departments represent ideal settings for vaccination efforts because each year millions of adults who have no or limited access to traditional primary care visit hospital EDs for medical and surgical problems that are non-life threatening. Such EDs often already provide other medical screening and preventive care services in the management of their patients. Almost one-quarter of adults aged 65 years and older make one or more visits to an emergency department each year. Patients who use EDs as their usual source of care are more likely to be members of minority groups and uninsured. These characteristics suggest that vaccination programs in EDs could have a significant impact in correcting disparities in vaccination coverage among patients in older age groups.

Combined with the large volume of patient visits each day, these characteristics would seem to make EDs ideal settings to implement vaccination services for people who have little access to primary care. Furthermore, influenza vaccination in EDs could play a substantial role in correcting disparities in vaccination coverage among this cohort of patients. The American College of Emergency Physicians recommends that ED personnel consider participating in influenza vaccine programs for the elderly if other sources of vaccination are not readily available.

A limited number of studies suggest that about half of patients for whom influenza vaccine is indicated (based on age or other high risk conditions) who have not yet received influenza vaccination during the current season would accept vaccination if it was offered to them during an ED visit. However, since these studies were conducted early in the vaccination season and involved the use of convenience samples, the results might not be generalizable to all patients seen in an ED throughout the vaccination season. The proportion of persons who would not have been vaccinated elsewhere but would accept vaccination in EDs has not been demonstrated. Therefore, the true potential of vaccination in EDs to increase vaccination coverage is unknown.

Additional evidence suggests that strong recommendation by a health care professional, particularly the patient's primary physician, can further increase the acceptance of influenza vaccine. However, there is limited evidence regarding the effectiveness of counseling by providers who are previously unknown to the patient, as is usually the case in an ED setting, to produce a similar change in patient behavior.

Goals and Objectives The overall goal is to determine the feasibility, sustainability, acceptability, and effectiveness of hospital-based vaccination efforts and to increase influenza immunization coverage among persons aged 18 years and older for whom vaccination is recommended who would otherwise not have been vaccinated. Inherent in feasibility and sustainability are the ability to recoup some income from those vaccinated.

Objective

For patients aged 18 years and older who seek medical care in the ED, determine

1. the number of vaccinations administered to eligible persons
2. the proportion of patients, among all persons not previously vaccinated, who accept vaccines in the emergency department.
3. the increase in coverage that can be achieved through a four-month emergency department-based vaccination program

Study design and methods

1. All patients aged 18 years and older will be approached by the PPS after the chief complaint is ascertained. The PPS will begin and administer a questionnaire on all eligible patients for whom vaccine is recommended. If the patient is eligible, the PPS will read the questionnaire to the patient.
2. If the patient is unsure or states that he or she does not want to receive the flu vaccine, the PPS will determine the reason for vaccine refusal.

If the patient meets criteria for influenza vaccination and/or pneumococcal vaccination, the PPS will inform him/her that influenza/pneumococcal vaccine is/are recommended for them and that the vaccination will be offered to eligible patients in the ED at no additional charge beyond that which is reimbursed by their insurance. Patients will be referred to a physician for additional assessment if they have a questionable or possible contraindication. The PPS will provide all eligible patients with the appropriate Vaccine Information Statement(s) and answer any questions. If the patient agrees to be vaccinated, the PPS will place a preprinted order form in the patient's chart, ask the physician to sign the order, and alert the patient's nurse. The patient will be offered vaccination by an ED nurse while they are undergoing evaluation and treatment in the emergency room. The nurse giving the vaccination will document the lot number, expiration date, time and location of the injection(s) on a label that will be placed in the patient's chart.

Documentation of doses received will be faxed to the patient's private care physician, if the information is available for doing so.

How confidentiality will be maintained:

Personal identifiers will not be retained by investigators beyond the time needed to document dose receipt in the patient medical record.

Exclusion criteria:

All patients under 18 years of age will be excluded. Any patient with a medically unstable condition, altered mental status, or language barrier will also be excluded. Patients who present with a contraindication to influenza vaccination (acute febrile illness or a history of allergic reaction to eggs) or pneumococcal vaccine will not be eligible for receipt of those vaccines.

Immunization status:

Previous immunization history will be assessed by patient self-report.

Data analysis:

The primary outcome measure will be the number of indicated influenza and pneumococcal vaccinations received during the course of the study. Data will be collected and analyzed according to demographic information, contraindications, and clinical consent.

PROTOCOL - Our Lady of the Lake Regional Medical Center

Goals and Objectives:

The overall goal is to determine the feasibility, sustainability, acceptability, and effectiveness of hospital-based vaccination efforts and to increase influenza immunization coverage among persons aged 50 years and older who would otherwise not have been vaccinated. Inherent in feasibility and sustainability are the ability to recoup some income from those vaccinated.

Objective

For patients aged 50 years and older who seek medical care in the ED, determine

1. the number of vaccinations administered
2. the proportion of patients, among all persons not previously vaccinated, who accept vaccines in the emergency department.
3. the increase in coverage that can be achieved through a four-month emergency department-based vaccination program
4. information or incentives that might convince initially reluctant patients to accept influenza vaccine

Study design and methods

1. All patients aged 50 years and older will be approached by the scribe after the chief complaint is ascertained. The scribe will begin and administer a questionnaire on all age eligible patients. Having already taken a history, the scribe will be able to easily determine if the patient is eligible for the study (i.e. does not meet any of the exclusion criteria). If the patient is eligible, the scribe will read the questionnaire to the patient.
2. If the patient is unsure or states that he or she does not want to be vaccinated, the scribe will determine the reason.

If the patient meets criteria for vaccination (i.e., has not been previously vaccinated against influenza this season and has no known contraindications to influenza vaccination), the scribe will inform him/her that influenza vaccine is recommended and that the vaccine will be offered to eligible patients in the ED at no additional charge beyond that which is reimbursed by their insurance. Patients will be referred to a physician for additional assessment if they have a questionable or possible contraindication. The scribe will provide all eligible patients with a VIS and answer any questions. If the patient agrees to be vaccinated, the scribe will place a preprinted label in the patient's chart, ask the physician to sign the order, and alert the patient's nurse. The patient will be offered vaccination by an ED nurse while they are undergoing evaluation and treatment in the emergency room. The nurse giving the vaccination will document the lot number, expiration date, time and location of the injection on a label that will be placed in the patient's chart.

How confidentiality will be maintained:

Personal identifiers will not be retained by investigators beyond the time needed to document dose receipt in the patient medical record.

Exclusion criteria:

All patients under 50 years of age will be excluded. Any patient with a medically unstable condition, altered mental status, or language barrier will also be excluded. Patients who present with a contraindication to influenza vaccination (acute febrile illness or a history of allergic reaction to eggs) or previous influenza vaccines will be excluded.

Immunization status:

Previous immunization history will be assessed by patient self-report.

Data analysis:

The primary outcome measure will be the number of indicated influenza vaccinations received during the course of the study. Data will be collected and analyzed according to demographic information, contraindications, and clinical consent.

Secondary analysis will be of the effectiveness of systems changes to deliver vaccine in an emergency department setting. If necessary, surveys will be administered to key staff persons to assist with data gathering for this analysis.

ELIGIBILITY:
Baton Rouge General Medical Center

Inclusion Criteria:

* Patients aged 18 years and older who are seeking medical care in the ED

Exclusion Criteria:

* All patients under 18 years of age will be excluded. Any patient with a medically unstable condition, altered mental status, or language barrier will also be excluded. Patients who present with a contraindication to influenza vaccination (acute febrile illness or a history of allergic reaction to eggs) or pneumococcal vaccine will not be eligible for receipt of those vaccines.

Our Lady of the Lake Regional Medical Center

Inclusion Criteria:

* Patients aged 50 years and older who are seeking medical care in the ED

Exclusion Criteria:

* All patients under 50 years of age will be excluded. Any patient with a medically unstable condition, altered mental status, or language barrier will also be excluded. Patients who present with a contraindication to influenza vaccination (acute febrile illness or a history of allergic reaction to eggs) or pneumococcal vaccine will not be eligible for receipt of those vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-12; Study Completion 2006-03

PRIMARY OUTCOMES:
Acceptance of vaccinations
Receipt of vaccination

SECONDARY OUTCOMES:
Reasons vaccines were refused
Reasons vaccines were not administered

CONTACTS AND LOCATIONS:
Overall Officials: William M Cassidy, MD, Principal Investigator — Louisiana State University Health Sciences Center; Daniel Fishbein, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana

REFERENCES:
- [Background] Harper SA, Fukuda K, Uyeki TM, Cox NJ, Bridges CB; Advisory Committee on Immunization Practices (ACIP), Centers for Disease Control and Prevention (CDC). Prevention and control of influenza. Recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2005 Jul 29;54(RR-8):1-40. PMID 16086456
- [Background] Centers for Disease Control and Prevention (CDC). Public health and aging: influenza vaccination coverage among adults aged > or =50 years and pneumococcal vaccination coverage among adults aged > or =65 years--United States, 2002. MMWR Morb Mortal Wkly Rep. 2003 Oct 17;52(41):987-92. PMID 14561957
- [Background] Pleis JR, Gentleman JF. Using the National Health Interview Survey: time trends in influenza vaccinations among targeted adults. Eff Clin Pract. 2002 May-Jun;5(3 Suppl):E3. PMID 12166924
- [Background] Ayanian JZ, Weissman JS, Schneider EC, Ginsburg JA, Zaslavsky AM. Unmet health needs of uninsured adults in the United States. JAMA. 2000 Oct 25;284(16):2061-9. doi: 10.1001/jama.284.16.2061. PMID 11042754
- [Background] U.S. Department of Health and Human Services: Office of Disease Prevention and Health Promotion--Healthy People 2010. Nasnewsletter. 2000 May;15(3):3. No abstract available. PMID 11987364
- [Background] Walls CA, Rhodes KV, Kennedy JJ. The emergency department as usual source of medical care: estimates from the 1998 National Health Interview Survey. Acad Emerg Med. 2002 Nov;9(11):1140-5. doi: 10.1111/j.1553-2712.2002.tb01568.x. PMID 12414462
- [Background] Polis MA, Smith JP, Sainer D, Brenneman MN, Kaslow RA. Prospects for an emergency department-based adult immunization program. Arch Intern Med. 1987 Nov;147(11):1999-2001. PMID 3675103
- [Background] Rodriguez RM, Baraff LJ. Emergency department immunization of the elderly with pneumococcal and influenza vaccines. Ann Emerg Med. 1993 Nov;22(11):1729-32. doi: 10.1016/s0196-0644(05)81313-7. PMID 8214864
- [Background] Slobodkin D, Zielske PG, Kitlas JL, McDermott MF, Miller S, Rydman R. Demonstration of the feasibility of emergency department immunization against influenza and pneumococcus. Ann Emerg Med. 1998 Nov;32(5):537-43. PMID 9795315
- [Background] Centers for Disease Control (CDC). Adult immunization: knowledge, attitudes, and practices--DeKalb and Fulton Counties, Georgia, 1988. MMWR Morb Mortal Wkly Rep. 1988 Nov 4;37(43):657-61. No abstract available. PMID 3141764
- [Background] Nicoleau A, Nicoleau CA, Balzora JD, Oboh A, Siddiqui N, Rosenberg C. Elderly African-Americans and the influenza vaccine: the impact of the primary care physician. J Am Med Dir Assoc. 2001 Mar-Apr;2(2):56-9. PMID 12812590
- [Background] National Center for Health Statistics (US). Health, United States, 2004: With Chartbook on Trends in the Health of Americans. Hyattsville (MD): National Center for Health Statistics (US); 2004 Sep. Report No.: 2004-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK20751/ PMID 20698065
- [Background] American College of Emergency Physicians. Immunization of adult patients. 2000. Ref Type: Report